CLINICAL TRIAL: NCT02679963
Title: A Randomized Double-blind Phase II Trial Evaluating Maintenance Olaparib Versus Placebo in Patients With Platinum-sensitive Advanced Non-small Cell Lung Cancer
Brief Title: Trial Evaluating Maintenance Olaparib in Patients With Platinum-sensitive Advanced Non-small Cell Lung Cancer
Acronym: PIPSeN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-005586-75; 2014/2204 (Other: CSET number)
Record Dates: First submitted 2016-01-26; First posted 2016-02-11 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maintenance Olaparib (Experimental): Olaparib (experimental arm): 600 mg daily (2 doses of 300 mg (2*2 tablets of 150 mg) taken approximately 12 hours apart) po, administered until disease progression or toxicity requiring its interruption. Olaparib has to be started no later than 6 weeks after the last administration of induction chemotherapy, and no later than 3 weeks after the CT scan confirming response to induction chemotherapy
  Interventions: Drug: Olaparib
- Placebo (Placebo Comparator): Placebo (control arm): 2 doses of 300 mg per day (2*2 tablets of 150 mg) taken approximately 12 hours apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olaparib
  Arms: Maintenance Olaparib
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multicentre randomised double-blind phase II trial, sponsored by Gustave Roussy and involving one French center as well as the Spanish Lung Cancer Group (≈20 centers of the SLCG).

Six hundred patients with diagnosis of stage IIIB/IV NSCLC will initially be registered prior to receiving the first line platinum-based chemotherapy or during or at the end of the first 6 cycles of inducation platinium based chemotherapy and provide consent for retrieving archival tissue collection and providing translational blood samples and tumor biopsies.

1. - Induction chemotherapy phase All patients will initially be treated with 6 cycles of platinum-based induction chemotherapy. Cycle duration will be 21 days. Doublets should either consist of a pemetrexed-platinum (cisplatin or carboplatin) doublet (preferentially for non-squamous NSCLC) or a gemcitabine - or vinorelbine - platinum doublet for squamous NSCLC. Taxanes-platinum doublets will not be accepted. Translational blood samples will be taken at the beginning of induction chemotherapy for all patients.

   Patients displaying progressive disease or stable disease after induction chemotherapy will be withdrawn and further optimally managed according to local practice. For them, an optional tumour biopsy will be performed at the end of the induction treatment.
2. - Randomisation and maintenance phase Only patients who respond to platinum-based induction chemotherapy will be further randomised between olaparib and placebo. These patients must have been treated with 6 cycles of chemotherapy. However, patients who haven't received 6 cycles of the induction chemotherapy due to severe toxicity (grade 3 or 4, NCI CTCAE v4.0) could be randomized only if they had received 4 chemotherapy cycles at least and if all treatment related toxicities are resolved to a grade ≤ 1 (NCI CTCAE v4.0).

Treatment will be administered at a dose of 600 mg daily (2 doses of 300 mg [2 tablets of 150 mg] taken approximately 12 hours apart) and cycle duration will be 28 days. Disease will be assessed every 2 cycles by CTscan (MRI or PET-scan if the scan is not contributive) and treatment will be administered until disease progression or unacceptable toxicity. Patients will then be optimally managed according to local practice. Follow-up will be for a minimum of 15 months from the time of randomization, and until last venue. All randomised patients will be asked to provide translational blood samples at randomization, on treatment and at the end of the treatment. Optional tumour biopsies will be performed at randomization, at the end of the treatment (or at disease progression if available).

ELIGIBILITY:
For inclusion in the study subjects should fulfill the following criteria:

1. Provision of written informed consent to treatment and companion translational studies prior to any study specific procedures
2. Patients must be > 18 years of age.
3. Affiliation to an health insurance
4. Histological diagnosis of NSCLC
5. Advanced or metastatic disease (stage IIIB/IV)
6. Access to the original tumor biopsy or planning of a fresh tumor biopsy before start the platinium based chemotherapy
7. Chemonaive for NSCLC or patient having received adjuvant chemotherapy at least 2 years before trial enrolment or patient currently receiving his/her first platinum-based chemotherapy for advanced NSCLC (first line or second line only if the first line was an anti-PD-1 or anti-PD-L1 agent monotherapy)
8. No other cancer in the previous 3 years, except cervical cancer or cutaneous cancer
9. Absence of EGFR-sensitising mutation or ALK translocation
10. ECOG Performance Status of 0-1
11. Fit to receive 6 cycles or currently receiving of platinum-based induction chemotherapy
12. At the start of the platinium based induction chemotherapy measurable lesions by RECIST v1.1 criteria, i.e. at least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10mm in the longest diameter (except lymph nodes that must have short axis ≥ 15mm) with computed tomography (CT), magnetic resonance imaging (MRI) or clinical examination and which is suitable for accurate repeated measurements.

    Inclusion criteria 13 is only for patients registered before starting the platinum-based induction chemotherapy:
13. Patients must have normal organ and bone marrow function measured within 14 days prior to administration of the platinum based treatment

    * Haemoglobin ≥ 10.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
    * Creatinine clearance > 60mL/min as calculated by Cockroft-Gault formula for cisplatin administration; creatinine clearance >/= 51mL/min by Cockroft-Gault formula for carboplatin administration
14. Evidence of non-childbearing status for women of childbearing potential: negative serum pregnancy test within 14 days of study treatment.

    Postmenopausal is defined as:
    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
    * LH and FSH levels in the post-menopausal range for women under 50,
    * Radiation-induced oophorectomy with last menses >1 year ago,
    * Chemotherapy-induced menopause with >1 year interval since last menses,
    * Or surgical sterilisation (bilateral oophorectomy or hysterectomy).
15. Both men and women (of childbearing potential) who are sexually active should accept to use adequate contraception, during and for at least 6 months post-treatment
16. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
17. Previous surgery (in the adjuvant setting) for NSCLC, radiotherapy (with a curative intent for local or locally-advanced disease) or immunotherapy by anti- PD-1 or anti-PD-L1 agent in the metastatic setting are allowed

Non-inclusion criteria:

1. Uncontrolled or symptomatic brain metastases. Controlled brain metastases are defined as stable for 1 month. A scan to confirm the absence of brain metastases is not required. Corticosteroids therapy will be allowed if administered at a stable dose for at least one month before entering the trial.
2. Previous enrolment (or randomisation) in the present study Any previous systemic treatment for cancer in the previous 3 years.
3. Any previous systemic treatment for cancer in the previous 3 years except for NSCLC.
4. Patients receiving any radiotherapy or considering to require radiotherapy to the lung at the time of study entry or in the near future, except for palliative reasons. The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to inclusion.
5. Patients receiving the following classes of inhibitors of CYP3A4 (see Section 6.5 for guidelines and wash out periods).

   * Azole antifungals
   * Macrolide antibiotics
   * Protease inhibitors
6. Major surgery within 14 days before to start the induction chemotherapy and patients who have not recovered from any effects of any major surgery.
7. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, coronary artery disease, cardiomyopathy, uncontrolled hypertension, myocardial infarction in the last 3 months, unstable spinal cord compression (untreated and unstable for at least 28 days prior to start the induction chemotherapy), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent.
8. Pregnant and/or breast-feeding women.
9. Patients who are known to be serologically positive for human immunodeficiency virus (HIV) and/or are receiving antiviral therapy. Systematic serologies to confirm the absence of this disease are not required.
10. Patients with known active hepatic disease (i.e., Hepatitis B or C) Systematic serologies to confirm the absence of these diseases are not required.
11. Patients with a known hypersensitivity to olaparib/placebo, cisplatin, carboplatin, or other platinum containing compounds, or any of the excipients of the product.
12. Concomitant yellow fever vaccine
13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of olaparib/placebo.
14. Symptomatic peripheral neuropathy ≥ grade 2
15. Patients with uncontrolled seizures
16. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
17. Enrolment in another clinical trial (except observational study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Assessed every 56 days up to 15 months
  By CT scan, MRI or TEP-scan according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Survival | Measured from patient randomization to death or last follow-up for patient alive or consent withdrawal up to 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus, Villejuif, Val de Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Postel-Vinay S, Coves J, Texier M, Aldea M, Gazzah A, Domine M, Planchard D, De Las Penas R, Sala Gonzalez MA, Viteri S, Perez J, Ortega AL, Moran T, Camps C, Lopez-Martin A, Provencio M, Soria JC, Besse B, Massuti B, Rosell R. Olaparib maintenance versus placebo in platinum-sensitive non-small cell lung cancer: the Phase 2 randomized PIPSeN trial. Br J Cancer. 2024 Feb;130(3):417-424. doi: 10.1038/s41416-023-02514-5. Epub 2023 Dec 14. PMID 38097741